CLINICAL TRIAL: NCT06701032
Title: Evolution of Hemodynamic Parameters in People With Atherosclerotic Vascular Disease Referred to a Secondary Prevention and Cardiovascular Rehabilitation (PREV) Program: a Prospective Cohort Study.
Brief Title: Hemodynamic Parameters in People With Atherosclerotic Vascular Disease Referred to a Secondary Prevention and Cardiovascular Rehabilitation Program
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: CISSS de Chaudière-Appalaches (Other Government)
Responsible Party: Principal Investigator, Jérôme Patry, Principal Investigator, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CISSSCA-2025-1208
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Peripheral Artery Disease (PAD); Coronary Artery Disease (CAD) (E.G., Angina, Myocardial Infarction, and Atherosclerotic Heart Disease (ASHD)); Cerebrovascular Atherosclerosis
Keywords: cardiovascular rehabilitation; supervised exercise therapy; secondary prevention; cardiovascular secondary prevention; cardiovascular rehabilitation program; hemodynamics of lower limbs; toe pressure measurement
MeSH Terms: conditions — Peripheral Arterial Disease; Coronary Artery Disease; Angina Pectoris; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cardiovascular rehabilitation program (Experimental)
  Interventions: Other: Cardiovascular rehabilitation program

INTERVENTIONS:
Other: Cardiovascular rehabilitation program — The cardiovascular rehabilitation program consists of a 12 weeks supervised exercises therapy (either in person or in tele-care)

SUMMARY:
The main purpose of this study is to evaluate the hemodynamic changes in the forefoot of patients with coronary, cerebrovascular or peripheral atherosclerotic disease referred a 12-week cardiovascular rehabilitation program (PREV program).

Also, this study will describe the characteristics of patients admitted to the PREV program and their evolutions in terms of favorable, unfavorable outcomes and complications and up to one year after completion of the program.

ELIGIBILITY:
Inclusion Criteria:

* Any individual aged 18 years and older who has been diagnosed with peripheral artery disease, coronary artery disease, angina, ischemic heart failure, transient ischemic attack or ischemic stroke (non-cardioembolic, non-hemorrhagic);
* Have been admitted to the PREV program;

Exclusion Criteria:

* Being not able to give written informed consent;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-08-29 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in toe pressure measurement | Change from baseline to 12 weeks
  Results will be measured in mm Hg
Change in the toe-brachial index | Change from baseline to 12 weeks
Change in the ankle-brachial index | Change from baseline to 12 weeks

SECONDARY OUTCOMES:
Change in 6-minute walk test (6MWT) | Change from Baseline to 12 weeks
  Results will be measured in meters
Short Form Health Survey 36 (SF-36) | Change from baseline to 12 weeks
  Change in quality of life measured using the SF-36 questionnaire. The scores range from 0-100.

CONTACTS AND LOCATIONS:
Locations (1):
- CLSC de Lévis - Programme PREV du CISSS de Chaudière-Appalaches, Lévis, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided